CLINICAL TRIAL: NCT03672591
Title: Cross-sectional Observational Single-center Study to Evaluate Renal Hemodynamics in Patients With Heart Failure and Preserved Ejection Fraction
Brief Title: Renal Hemodynamics in Patients With HFpEF
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Principal Investigator, Roland E. Schmieder, Head of the Clinical Research Center, University of Erlangen-Nürnberg Medical School
Other Study IDs: CRC2018HFpEF
Record Dates: First submitted 2018-09-04; First posted 2018-09-14 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure With Normal Ejection Fraction
Keywords: Heart failure; Renal clearance technique; Preserved ejection fraction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — * Biochemistry (urea, serum creatinine, eGFR, cystatin C, uric acid, sodium, potassium, calcium, phosphate, lipid levels, total protein, SGOT, SGPT, AP, ɣ-GT)
  * Hematology (hemoglobin, hematocrit, red blood cell count, platelet count, white blood cell count)
  * Fasting blood glucose, HbA1c
  * NT-proBNP
  * TSH
  * Spot-urine (urinary creatinine and albumin, urinary sodium and potassium)
  * Urinary dip stick analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HFpEF patients: Patients suffering from heart failure with preserved ejection fraction
  Interventions: Other: Renal clearance examination
- Control group: Subjects without HFpEF who participated in different studies during which renal clearance examination has been performed with the constant infusion input clearance technique in our Clinical Research Center (clin. gov. numbers: NCT00627952, NCT01835678, NCT00136188, NCT00905528, NCT00160745)
  Interventions: Other: Renal clearance examination

INTERVENTIONS:
Other: Renal clearance examination — Evaluation of renal hemodynamic parameters by constant-infusion input clearance technique with p-aminohippuric acid and Iohexol
  Other Names: Scanning laser Doppler flowmetry, SphygmoCor, UnexEF

SUMMARY:
Impaired renal function and heart failure with preserved ejection fraction (HFpEF) are two often co-existing medical conditions and are known to be associated with adverse cardiovascular outcome and increased mortality. The relationship between HFpEF and renal impairment is bidirectional. On the one hand, renal dysfunction has been shown to be an independent risk factor for the development of HFpEF. On the other hand, an increase in central venous pressure leading to renal dysfunction by a reduction of renal blood flow (RBF) and perfusion pressure (RPP) as well as activation of the renin-angiotensin-aldosterone system (RAAS) in patients with HFpEF has been previously described.

In the literature, several studies aimed to investigate the association between renal (dys-) function and HFpEF. In all these studies, renal function was assessed by determination of standard kidney function parameters such as serum creatinine, eGFR and urinary albumin to creatinine ratio (UACR). Constant infusion input clearance technique however offers a more detailed evaluation of renal function and hemodynamics. To the best of knowledge, renal hemodynamics in patients with HFpEF have not yet been investigated by clearance technique. Therefore, the aim of the present study is to evaluate renal function and hemodynamics by means of constant infusion input clearance technique with sodium p-aminohippuric acid (PAH) and Iohexol in 40 patients with HFpEF. The constant infusion input clearance technique offers an exact evaluation of renal function by measuring (not estimating) glomerular filtration rate and renal hemodynamic parameters such as renal plasma flow (RPF), filtration fraction (FF) and intraglomerular pressure (IGP). These results will be compared to 140 subjects without HFpEF that have participated in various studies and have been analyzed with the same constant infusion input clearance technique performed in the Clinical Research Center of the University Hospital Erlangen-Nuremberg. Additionally, flow mediated vasodilation (FMD), pulse wave velocity and parameters of retinal vascular remodeling by means of scanning laser Doppler flowmetry (SLDF) will be assessed in patients with HFpEF thereby allowing to examine the relationship between vascular remodeling in the systemic and renal circulation.

DETAILED DESCRIPTION:
Several studies evaluating the outcome among patients with HFpEF revealed that this entity of heart failure (HF) is associated with high mortality rates and some studies even indicate that mortality is similar to patients with heart failure and reduced ejection fraction (HFrEF). Hospitalization for HFpEF is increasing relative to HFrEF, highlighting the need for a better understanding of the pathogenetic processes in order to develop new treatment strategies for this type of HF. Recently, the PARAMOUNT study revealed that in patients with HFpEF, treatment with the dual-acting angiotensin receptor neprilysin inhibitor (ARNI) LCZ696 was associated with lower levels of creatinine and higher estimated glomerular filtration rates (eGFR) indicating a better preservation of renal function in comparison to treatment with valsartan only. Another observation of this study was an increase in urinary albumin to creatinine ratio (UACR) in the group of LCZ696-treatment, which was not visible in patients randomized to the valsartan group. Additionally, analysis of the relation between albuminuria and/or decreased eGFR and cardiovascular function and structure revealed that renal dysfunction was common in this group of patients and associated with cardiac remodeling and dysfunction.

Up to two thirds of patients with HFpEF are suffering from chronic kidney disease (CKD). A bidirectional cardiorenal relation has been recently described and is known to be associated with adverse cardiovascular outcome and increased mortality. On the one hand, renal dysfunction has been shown to be an independent risk factor for the development of HFpEF due to inflammatory processes and endothelial dysfunction. On the other hand, an increase in central venous pressure leading to renal dysfunction by a reduction of renal blood flow (RBF) and perfusion pressure (RPP) as well as activation of the renin-angiotensin-aldosterone system (RAAS) in patients with HFpEF has been previously described.

This association has also been demonstrated for patients with HFrEF. However, several studies comparing patients with the two subtypes of HF in the context of CKD indicate that this association is more pronounced in patients with HFpEF. For example, a community-based cohort study by Brouwers et al. including 8592 subjects of the PREVEND trial showed that renal function parameters such as urinary albumin excretion (UAE) and cystatin C were associated with a high risk for the development of HFpEF but not HFrEF. Ahmed et al. even reported a higher CKD-related mortality in HFpEF than in HFrEF patients with an underlying graded-response relation as CKD-associated mortality increased with higher left ventricular ejection fraction (LVEF). These findings suggest different pathogenetic processes for these two subtypes of HF. Therefore, detailed exploration of the pathophysiological mechanisms behind the relationship of HFpEF and renal function represents a matter of major research interest.

Recently, several studies aimed to investigate the association between renal (dys-) function and HFpEF. Unger et al. retrospectively examined the relationship between renal function and echocardiographic parameters in 299 patients with HFpEF. The analysis revealed that CKD was independently associated with worse cardiac mechanics and outcomes in this population.9 Studying 217 participants from the PARAMOUNT trial with HFpEF, Gori et al. demonstrated that renal dysfunction was associated with abnormal left ventricular geometry, lower midwall fractional shortening and higher NT-proBNP. In both studies, renal function was assessed with commonly used tests such as determination of serum creatinine, eGFR and urinary albumin to creatinine ratio (UACR). However, these parameters only allow an approximate estimation of renal function. Constant infusion input clearance technique offers a more complete approach towards evaluation of renal function and perfusion, allowing an exact quantification of glomerular filtration rate (GFR) and renal hemodynamic parameters such as renal plasma flow (RPF), filtration fraction (FF) and intraglomerular hemodynamics.

The definition of HFpEF in literature is rather inconsistent. In some studies, HFpEF was defined by an ejection fraction of ≥ 45%, whereas other authors used a cut-off value of 50%. In the present study, the categorization of heart failure as HFpEF will follow the 2016 European Society of Cardiology (ESC) guidelines for the diagnosis and treatment of acute and chronic heart failure applying a cut-off value of 50%.

The purpose of the present study is to evaluate renal function and hemodynamics by means of constant infusion input clearance technique with PAH and Iohexol in 40 patients with HFpEF with the aim to better characterize the relationship between renal dysfunction and HFpEF. These results will be compared to 140 subjects without HFpEF who participated in different studies during which renal clearance examination has been performed with the constant infusion input clearance technique in the Clinical Research Center of the University Hospital Erlangen-Nuremberg. In parallel, pulse wave velocity, flow mediated vasodilation and other vascular parameters, reflecting the vascular wall properties of small and large arteries, will be assessed. Additionally, there will be a non-invasive retinal examination to assess vascular remodeling of retinal arterioles (wall to lumen ratio, WLR), retinal capillary flow (RCF) and capillary rarefaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients in good and stable health condition
* Informed consent has to be given in written form
* HFpEF in stable conditions according to 2016 ESC guidelines definition14

  * LVEF ≥ 50%
  * symptoms and/or signs of CHF
  * NT-proBNP > 125 pg/ml
  * At least one additional criterion: relevant structural heart disease (left ventricular hypertrophy and/or left atrial enlargement and/or diastolic dysfunction

Exclusion Criteria:

* Uncontrolled diabetes (fasting plasma glucose ≥ 240 mg/dl, HbA1c ≥ 10%)
* Uncontrolled arterial hypertension (≥ 180/110 mmHg)
* Any history of stroke, transient ischemic attack, instable angina pectoris or myocardial infarction within the last 6 months prior to study inclusion
* Significant valvular heart disease
* Known hypertrophic obstructive cardiomyopathy or known pericardial constriction
* Atrial fibrillation with a resting heart rate > 90 bpm
* Heart transplant recipient
* Sickle cell anemia
* Pheochromocytoma
* Myasthenia gravis
* Subclinical or clinical hyperthyroidism
* Allergic reaction to iodine
* Medication with amiodarone
* Estimated glomerular filtration rate < 30 ml/min/1.73m²
* Significant laboratory abnormalities such as Serum Glutamate-Oxaloacetate-Transaminase (SGOT) or Serum Glutamate-Pyruvate-Transaminase (SGPT) levels more than 3 times above the upper limit of normal range
* Patients in unstable conditions due to any kind of serious disease, that infers with the conduction of the trial
* History of epilepsia and history of seizures
* Patients suffering from cataract or glaucoma
* Diabetic retinopathy
* Drug or alcohol abuse
* Pregnant and breast-feeding patients
* Body mass index > 40 kg/m²
* Participation in another clinical study within 30 days prior to visit 1
* Individuals at risk for poor protocol adherence
* Subjects who do not give written consent, that pseudonymous data will be transferred in line with the duty of documentation and the duty of notification according to § 12 and § 13 GCP-V

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HFpEF patients: recruitment from the investigator's outpatient clinics and referring physicians.
  Control subjects without HFpEF: individuals who already participated in different studies during which renal clearance examination has been performed with the constant infusion input clearance technique in our Clinical Research Center (clin. gov. numbers: NCT00627952, NCT01835678, NCT00136188, NCT00905528, NCT00160745)
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Renal plasma flow | One week after study inclusion
  Volume of blood plasma delivered to the kidneys per unit time (ml/min)

SECONDARY OUTCOMES:
Flow mediated vasodilation | One week after study inclusion
  Measured by UNEX EF in percent
Wall to lumen ratio of retinal arterioles | One week after study inclusion
  ratio of vascular wall thickness to luminal diameter
Retinal capillary flow | One week after study inclusion
  by SLDF measurement in AU
Office and 24-hour systolic, diastolic and mean ambulatory blood pressure | One week after study inclusion
  in mmHg
Central systolic pressure | One week after study inclusion
  measured by SphygmoCor in mmHg
Pulse pressure | One week after study inclusion
  difference between systolic and diastolic blood pressure in mmHg
Pulse wave velocity | One week after study inclusion
  velocity at which the blood pressure pulse propagates through the circulatory System measured by SphygmoCor in m/s
Glomerular filtration rate | One week after study inclusion
  Flow rate of filtered fluid through the kidney in ml/min/1.73m^2
Filtration fraction | One week after study inclusion
  Ratio of glomerular filtration rate to renal plasma flow in percent
Renal vascular resistance | One week after study inclusion
  Calculated by the Gomez formula in dyn x sec x cm^-5
Intraglomerular pressure | One week after study inclusion
  in mmHg

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Clinical Research Center Erlangen, Department of Nephrology and Hypertension, University Hospital Erlangen, Erlangen
  - Clinical Research Center Nuremberg, Department of Nephrology, University Hospital Erlangen, Nuremberg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jung S, Bosch A, Kolwelter J, Striepe K, Kannenkeril D, Schuster T, Ott C, Achenbach S, Schmieder RE. Renal and intraglomerular haemodynamics in chronic heart failure with preserved and reduced ejection fraction. ESC Heart Fail. 2021 Apr;8(2):1562-1570. doi: 10.1002/ehf2.13257. Epub 2021 Feb 9. PMID 33559346